CLINICAL TRIAL: NCT00500448
Title: The Efficacy of Neuromuscular Electrical Stimulation for Improving Quadriceps Activation in Women With Medial Tibiofemoral Osteoarthritis
Brief Title: An Intervention of Electrical Stimulation in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Palmieri-Smith
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis
Keywords: Arthritis, Knee, Quadriceps, Electrical Stimulation, Women
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Treatment (No Intervention): No treatment was delivered to this arm. Participants went about activities of daily living
- Electrical Stimulation (Experimental): Neuromuscular electrical stimulation treatments 3 times per week for 4 weeks
  Interventions: Device: Electrical Stimulation

INTERVENTIONS:
Device: Electrical Stimulation — Electrical Stimulation (NMES) will be delivered 3 times per week for 4 weeks
  Other Names: Vectra Genisys
  Arms: Electrical Stimulation

SUMMARY:
Patients with knee osteoarthritis (OA) often have decreased thigh muscle strength. This muscle weakness is thought to originate from centers in the brain and spinal cord that restrict recruitment of fibers responsible for muscle contraction. An inability to fully contract muscles surrounding the knee joint impairs patients' abilities to perform activities of daily living (i.e. walking, climbing stairs) and may even contribute to further joint degeneration.

Establishing therapies aimed at increasing muscle strength, restoring normal function, and possibly slowing the processes involved in the development of knee OA is essential in order to enhance the quality of life in the adult population plagued with this degenerative joint condition.

Electrical muscle stimulation applied to the thigh is a promising therapy that has been shown to successfully restore muscle strength, however how long the treatment lasts and its influence on functional outcomes remains unknown. In order for electrical muscle stimulation to be of value it must result in sustained improvements in muscle strength and functional outcomes. Therefore, the purpose of the proposed investigation is to determine if electrical muscle stimulation can restore thigh muscle strength and improve functional outcomes in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
A frequent clinical obstacle encountered in patients with knee osteoarthritis (OA) is an inability to achieve full voluntary activation of the quadriceps musculature. This phenomenon has been termed arthrogenic muscle inhibition (AMI) and is an ongoing reflex inhibition of musculature surrounding a joint following distension or damage to the structures of that joint. AMI is a limiting factor in joint rehabilitation as it restricts full muscle activation and therefore prevents restoration of strength. Thus, patients often participate in life activities deficient in strength and neuromuscular control resulting in altered lower extremity mechanics and potentially predisposing patients to further joint degeneration. Neuromuscular electrical stimulation (NMES) has been shown to be successful in reversing quadriceps AMI, however the duration of its effectiveness and its influence on functional outcomes remains elusive. Therefore, the purpose of the proposed study is to examine quadriceps activation and functional outcomes following a 4-week NMES protocol in patients with medial tibiofemoral osteoarthritis. To examine the efficacy of NMES in reversing AMI and improving functional outcomes, 38 subjects will be randomly assigned to either undergo a 4-week NMES program or to undergo no therapeutic intervention. Prior to treatment and at 1, 12, and 24 weeks following treatment, patients' quadriceps central activation ratios will be assessed. Additionally, subjects will undergo gait and stair climb analyses to determine if functional performance during these activities of daily living are improved when compared to the baseline assessment. Patients' perceived level of function will also be tested using the Western Ontario and McMasters Universities Osteoarthritis Index.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be female
* Subjects must have radiographic osteoarthritis of grade 2 severity according to the Kellgren and Lawrence scale on the posterior-anterior semi-flexed view with definite osteophytes present in the medial and not lateral compartment.

Exclusion Criteria:

* Previous adverse reaction to electrical stimulation
* Inability to ambulate without the use of an assistive device (i.e cane, walker)
* Patients who have undergone a total knee arthroplasty
* Patients who have torn any knee ligament (ACL, PCL, MCL, LCL)
* Enrollees who have a demand-type cardiac pacemaker or are pregnant
* History of tibial osteotomy surgery
* Significant peripheral or central nervous system disease
* Concurrent clinically active arthritis of the hip, ankle, hindfoot or midfoot in either limb
* Concurrent bilateral radiographic evidence of tibiofemoral osteoarthritis
* Enrollees who are concurrently undergoing physical therapy for pain or OA
* Enrollees who are taking Cox-2 inhibitors or are receiving corticosteroid injections
* Subjects will be allowed to take buffered aspirin and naproxen sodium while enrolled in the study
* Enrollees who have a body mass index of greater than 40 (morbidly obese)
* Enrollees who have a CAR > .95 (e.g. patients whose quadriceps are uninhibited)
* Enrollees who have previously undergone quadriceps NMES therapy

Ages: 50 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riann M Palmieri-Smith, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Palmieri-Smith RM, Thomas AC, Karvonen-Gutierrez C, Sowers M. A clinical trial of neuromuscular electrical stimulation in improving quadriceps muscle strength and activation among women with mild and moderate osteoarthritis. Phys Ther. 2010 Oct;90(10):1441-52. doi: 10.2522/ptj.20090330. Epub 2010 Jul 29. PMID 20671100

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuromuscular Electrical Stimulation: Neuromuscular electrical stimulation treatments 3 times per week for 4 weeks
  Neuromuscular Electrical Stimulation (Vectra Genisys 4 Channel Electrotherapy System): Estim will be delivered 3 times per week for 4 weeks
Period: Overall Study
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (2.9) | 58 (2.7) | 57.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Height [Mean (Standard Deviation); unit: cm] | 163.3 (4.5) | 162.3 (7.4) | 162.8 (5.95)
Mass [Mean (Standard Deviation); unit: kg] | 87.8 (12.5) | 86.3 (13.6) | 87.05 (13.05)
BMI [Mean (Standard Deviation); unit: kg^m2] | 32.1 (5.1) | 32.7 (4.1) | 32.4 (4.6)
Quadriceps Strength [Mean (Standard Deviation); unit: Nm/kg] | 1.24 (0.35) | 1.29 (0.46) | 1.26 (0.41)
Central Activation Ratio (CAR) [Mean (Standard Deviation); unit: ratio] — Knee extensionTorque recorded during voluntary contraction/Knee extension torque recorded during contraction with superimposed stimulus
  ratio | .83 (.15) | .90 (.08) | .86 (.12)
WOMAC Pain Score [Mean (Standard Deviation); unit: units on a scale (range 5-25)] — WOMAC Pain Score ranges from 5 (no pain) to 25 (worst possible pain)
  units on a scale (range 5-25) | 8.9 (4.3) | 7.6 (2.7) | 8.25 (3.5)
WOMAC disability scale [Mean (Standard Deviation); unit: units on a scale (range 17-85)] — WOMAC Disability Score ranges from 17 (no loss of function) to 85 (severe loss of function)
  units on a scale (range 17-85) | 28.8 (15.3) | 27.1 (12.1) | 27.95 (13.7)
Timed Walking speed [Mean (Standard Deviation); unit: m/s] | 1.40 (.13) | 1.43 (.19) | 1.42 (.16)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quadriceps Central Activation Ratio at 12 Weeks
Description: Knee extension Torque recorded during voluntary contraction/Knee extension torque recorded during contraction with superimposed stimulus
Time Frame: Baseline and 12 weeks post-intervention
Measure: Mean (95% Confidence Interval); unit: unitless
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 14 | 16
unitless | 0.01 [-0.09 to 0.10] | -0.04 [-.11 to 0.03]

2. Secondary Outcome: Change From Baseline in WOMAC Disability Score at 12 Weeks
Description: Womac Disability Score is on a scale from 17 (no functional loss) to 85 (severe functional loss)
Time Frame: baseline and 12 weeks post-intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 14 | 15
units on a scale | 5.0 [.59 to 9.41] | -4.92 [-10.89 to 1.05]

3. Secondary Outcome: Change From Baseline in Timed Walking Speed at 12 Weeks
Time Frame: Baseline and 12 weeks post-intervention
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 14 | 16
m/s | 0.04 [-0.09 to 0.17] | -0.05 [-0.13 to 0.03]

4. Secondary Outcome: Change From Baseline in WOMAC Pain Score at 12 Weeks
Description: WOMAC Pain Score ranges from 5 (no pain) to 25 (worst possible pain)
Time Frame: Baseline and 12 weeks following intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 14 | 16
units on a scale | 1.4 [-0.26 to 3.06] | -0.54 [-1.83 to 0.75]

5. Primary Outcome: Change From Baseline in Quadriceps Strength at 12 Weeks
Time Frame: Baseline and 12 weeks following the intervention
Measure: Mean (95% Confidence Interval); unit: Nm/kg
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 14 | 16
Nm/kg | .14 [-.20 to 0.49] | -0.21 [-0.50 to 0.08]

ADVERSE EVENTS:
Arm/Group | No Treatment | Neuromuscular Electrical Stimulation
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No